CLINICAL TRIAL: NCT02555371
Title: A Multi-center, Randomized, Double-blind, Placebo Controlled, Parallel Group Study to Compare Cessation Versus Continuation of Long-term Mepolizumab Treatment in Patients With Severe Eosinophilic Asthma (201810)
Brief Title: Cessation Versus Continuation of Long-term Mepolizumab in Severe Eosinophilic Asthma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201810; 2015-002361-32 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Asthma
Keywords: Severe eosinophilic asthma; mepolizumab; asthma exacerbation
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm Mepolizumab 100 mg (Experimental): There will be 4 parts during the study. Part A will be Variable Open-Label Run-in (maximum up to 132 weeks). Part B- Fixed Open-Label Run-In (4 Weeks to 8 weeks). Part C will be randomized double-blind treatment period (Up to 52 weeks) and in case of clinically significant asthma exacerbation, optional open label switch Part D (Up to 52 weeks post randomization). Subjects will receive mepolizumab (100 mg SC) every 4 weeks throughout study
  Interventions: Biological: Mepolizumab 100mg
- Arm Placebo (Placebo Comparator): There will be 4 parts during the study. Part A will be Variable Open-Label Run-in (maximum up to 132 weeks). Part B- Fixed Open-Label Run-In (4 Weeks to 8 weeks). Part C will be randomized double-blind treatment period (Up to 52 weeks) and in case of clinically significant asthma exacerbation, optional open label switch Part D (Up to 52 weeks post randomization). During Part A, B and D, subjects will receive open label mepolizumab (100 mg SC) every 4 weeks and during Part C, subjects will receive placebo SC every 4 weeks.
  Interventions: Biological: Mepolizumab 100mg; Drug: Placebo

INTERVENTIONS:
Biological: Mepolizumab 100mg — Mepolizumab is a fully humanised Immunoglobulin (IgG) antibody (IgG1, kappa) with human heavy and light chain frameworks. Mepolizumab will be provided as a lyophilised cake in sterile vials for individual use.
Drug: Placebo — The placebo will be 0.9% sodium chloride solution and will be provided by the study site.
  Arms: Arm Placebo

SUMMARY:
Primary objective of the study is to evaluate whether patients with severe eosinophilic asthma who have received long-term treatment with mepolizumab (at least 3 years) need to maintain treatment with mepolizumab to continue to receive benefit. Subjects who participated in the open-label studies MEA115666 or 201312 with at least 6 months of treatment with mepolizumab prior to Visit 1 and who have no more than 2 consecutive missed doses of mepolizumab treatment will be eligible to participate in this study. This study will be conducted in 4 parts in approximately 300 subjects. Part A will be Variable Open-Label Run-in (for subjects with less than 3 years of mepolizumab treatment). Once the required 3 year exposure is reached, subjects will enter Part B- Fixed Open-Label Run-In (4 weeks to 8 weeks). During Part A and B subjects will be administered Open-label mepolizumab (100 milligram [mg] Subcutaneous [SC]) every 4 weeks. Part C will be the randomized double-blinded part. Upon completion of Part B, eligible subjects will be randomized to mepolizumab (100 mg SC) every 4 weeks or placebo administered SC every 4 weeks for 52 weeks.

Subjects discontinuing investigational product (IP) due to a clinically significant asthma exacerbation will then enter optional Part D of the study. During Part D, subjects receive open-label mepolizumab in addition to their standard of care therapy for the remainder of the study, through Part D up to 52-weeks post-randomization. An Exit Visit will be conducted 52 weeks after randomization in order to assess subject's efficacy parameters, immunogenicity status, and to conduct additional safety assessments. Eligible subjects will participate in the study ranging from 56 to192 weeks, depending on the duration of Part A (0 to 132 weeks) and Part B (4 to 8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: Prior to commencing any study related activities, subjects must be able and willing to provide written informed consent, and an assent for subjects under 18 years of age, at Visit 0 (or Visit 1 if these Visits are conducted on the same day).
* MEA115666 or 201312 Study Participation: Participation (through the Follow Up/Exit Visit or Early Withdrawal) in either study with documented evidence of at least 6 months of continuous mepolizumab treatment prior to Visit 1. Continuous treatment with mepolizumab is defined as no more than 2 consecutive missed doses (no treatment gaps of more than 12 weeks [84 days] between any two doses).
* Current Anti-Asthma Therapy: Asthma is currently being treated with a controller medication and the subject has been on a controller medication for the past 12 weeks. Subjects will be expected to continue controller therapy for the duration of the study.
* Male or Eligible Female Subjects: A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, > 45 years, in the absence of hormone replacement therapy.

OR Child bearing potential, has a negative pregnancy test at screening, and agrees to acceptable contraceptive methods approved in their local country, when used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician) for the duration of the study and for 4 months after the last study drug administration.

A urine pregnancy test is required of all females of child-bearing potential at each scheduled study visit prior to the injection of study treatment, and at the Exit Visit, Early Withdrawal (EW) or Discontinuation of IP Visit.

* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* MEA115666 or 201312 IP Discontinuation: Subjects withdrawn from IP or withdrawn from study participation from either MEA115666 or 201312 for safety reasons.
* Health Status: Clinically significant deterioration in health status at the completion of participation or EW from either the MEA115666 or 201312 trials which in the opinion of the investigator would make the subject unsuitable for participation in this study.
* Pregnancy: Subjects who are pregnant or breastfeeding. Subjects should not be enrolled if they plan to become pregnant during the time of study participation.
* Cardiovascular: Subjects who have severe or clinically significant cardiovascular disease uncontrolled with standard treatment. Including but not limited to:

known ejection fraction of <30% OR severe heart failure meeting New York Heart Association Class IV classification OR hospitalised in the 12 months prior to Visit 1 for severe heart failure meeting New York Heart Association Class III OR angina diagnosed less than 3 months prior to Visit 1 or at Visit 1.

* 12-Lead Electrocardiogram (ECG): ECG which has a clinically significant abnormality observed at the Screening Visit as determined by the investigator. Subjects with the following abnormalities are excluded from study participation: QT interval corrected for heart rate by Fridericia's formula (QTcF) > 450 milliseconds (msec), or QTcF >480 msec for subjects with Bundle Branch Block.
* Malignancy: A current malignancy or previous history of cancer in remission for less than 12 months prior to screening (Subjects that had localized carcinoma of the skin which was resected for cure will not be excluded).

Note for South Korea: Korean subjects with a diagnosis of malignancy within 5 years are excluded.

* Other Monoclonal Antibodies: Subjects who have received any monoclonal antibody (other than XOLAIR®) to treat inflammatory disease within 5 half-lives of Visit 1.

XOLAIR is a registered trademark of Genentech USA, Inc. and Novartis Pharmaceuticals Corporation.

* Adherence: Subjects who have known evidence of lack of adherence within studies MEA115666 or 201312 (less than 80%) to controller medications, scheduled study visits and/or ability to follow physician's recommendations.
* Smoking status: Current smokers
* Inability to read: In the opinion of the Investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (66):
- United States (13):
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Murray, Utah
- Argentina (4):
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
- Australia (2):
  - GSK Investigational Site, New Lambton, New South Wales
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (3):
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Québec
- France (5):
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Paris
- Germany (6):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Magdeburg
- Japan (7):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Leeuwarden
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Wroclaw
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
- Russia (4):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Korea (6):
  - GSK Investigational Site, Anyang-Si, Gyeonggi-do
  - GSK Investigational Site, Bucheon-si, Gyeonggi-do
  - GSK Investigational Site, Cheongju-si, Chungcheongbuk-do
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon-si, Gyeonggi-do
- Spain (4):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Sabadell (Barcelona)
- Ukraine (4):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Mykolayiv
  - GSK Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Moore WC, Kornmann O, Humbert M, Poirier C, Bel EH, Kaneko N, Smith SG, Martin N, Gilson MJ, Price RG, Bradford ES, Liu MC. Stopping versus continuing long-term mepolizumab treatment in severe eosinophilic asthma (COMET study). Eur Respir J. 2022 Jan 6;59(1):2100396. doi: 10.1183/13993003.00396-2021. Print 2022 Jan. PMID 34172470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center, randomized, double-blind, placebo controlled, parallel group study to compare cessation versus continuation of long-term mepolizumab treatment. Participants (par.) who completed the Follow Up/Exit Visit or Early Withdrawal Visit from study MEA115666 (NCT01691859) or 201312 (NCT02135692) were eligible to participate in this study.
Pre-assignment Details: This is a 3 period study including variable open-label (OL) run-in, double-blind (DB) treatment period and open-label treatment switch period. The study was conducted in 75 centers across 14 countries from 07-Jan-2016 to 24-Jul-2019.
Groups:
- Part A/B: Mepolizumab 100mg SC: Participants with less than 3 years of mepolizumab treatment entered variable open-label run-in period-Part A in order to reach 3 years of exposure and received 100 mg of mepolizumab injected subcutaneously (SC) once every 4 weeks (W) up to 132 weeks. Upon achieving 3 years exposure, participants entered Part B. Participants with at least 3 years of mepolizumab treatment directly entered fixed open-label run-in period-Part B and received 100 mg of mepolizumab injected SC once every 4 weeks up to 8 weeks.
- Part C: Placebo: Upon completion of the fixed run-in period, participants entered a double-blind study treatment and received placebo SC every 4 weeks up to 52 weeks. Participants who experienced a clinically significant asthma exacerbation were assessed by the investigator to determine if they could continue double-blind treatment or should instead enter OL mepolizumab 100 mg SC every 4 weeks for the remainder of the treatment period (up to 52 weeks post-randomization).
- Part C: Mepolizumab 100mg SC: Upon completion of the fixed run-in period, participants entered a double-blind study treatment and received continued mepolizumab 100 mg SC every 4 weeks up to 52 weeks. Participants who experienced a clinically significant asthma exacerbation were assessed by the investigator to determine if they could continue double-blind treatment or should instead enter OL mepolizumab 100 mg SC every 4 weeks for the remainder of the treatment period (up to 52 weeks post-randomization).
- Part D: Mepolizumab 100mg SC (Previous Placebo): Participants who experienced a clinically significant asthma exacerbation were assessed by the investigator to determine if they could continue double-blind treatment or should instead enter OL mepolizumab 100 mg SC every 4 weeks for the remainder of the treatment period (up to 52 weeks post-randomization in Part C).
- Part D: Mepolizumab 100mg SC (Previous Mepolizumab): Participants who experienced a clinically significant asthma exacerbation were assessed by the investigator to determine if they could continue double-blind treatment or should instead enter OL mepolizumab 100 mg SC every 4 weeks for the remainder of the treatment period (up to 52 weeks post-randomization in Part C ).
Period: PartA(Upto 132W)+PartB(Upto 8W)
Arm/Group | Part A/B: Mepolizumab 100mg SC | Part C: Placebo | Part C: Mepolizumab 100mg SC | Part D: Mepolizumab 100mg SC (Previous Placebo) | Part D: Mepolizumab 100mg SC (Previous Mepolizumab)
Started (Variable & fixed run-in periods have been combined since all par. received OL mepolizumab 100 mg SC) | 306 | 0 | 0 | 0 | 0
Completed | 295 | 0 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Failure to meet continuation criteria | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 0
Period: Part C (DB Period: Up to 52W)
Arm/Group | Part A/B: Mepolizumab 100mg SC | Part C: Placebo | Part C: Mepolizumab 100mg SC | Part D: Mepolizumab 100mg SC (Previous Placebo) | Part D: Mepolizumab 100mg SC (Previous Mepolizumab)
Started (Double-blind Treatment Period) | 0 | 151 | 144 | 0 | 0
Completed | 0 | 62 | 96 | 0 | 0
Not Completed | 0 | 89 | 48 | 0 | 0
Not completed — Switched to Part D treatment | 0 | 84 | 45 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 1 | 0 | 0
Period: PartD(OL: 52W Post-randomization PartC)
Arm/Group | Part A/B: Mepolizumab 100mg SC | Part C: Placebo | Part C: Mepolizumab 100mg SC | Part D: Mepolizumab 100mg SC (Previous Placebo) | Part D: Mepolizumab 100mg SC (Previous Mepolizumab)
Started | 0 | 0 | 0 | 84 | 45
Completed | 0 | 0 | 0 | 80 | 42
Not Completed | 0 | 0 | 0 | 4 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Parts A/B: Mepolizumab 100mg SC: Participants with less than 3 years of mepolizumab treatment entered variable open-label run-in period-Part A in order to reach 3 years of exposure and received 100 mg of mepolizumab injected subcutaneously (SC) once every 4 weeks up to 132 weeks. Upon achieving 3 years exposure, participants entered Part B. Participants with at least 3 years of mepolizumab treatment directly entered fixed open-label run-in period-Part B and received 100 mg of mepolizumab injected SC once every 4 weeks up to 8 weeks.
Arm/Group | Parts A/B: Mepolizumab 100mg SC
Number analyzed (Participants) | 306
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180
  Male | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - CENTRAL/SOUTH ASIAN HERITAGE | 1
  ASIAN - EAST ASIAN HERITAGE | 28
  ASIAN - JAPANESE HERITAGE | 21
  BLACK OR AFRICAN AMERICAN | 8
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 3
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 245

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With First Clinically Significant Exacerbation in Part C
Description: Clinically significant exacerbation was defined as worsening of asthma which requires use of systemic corticosteroids (e.g., prednisone) for at least 3 days or a single intramuscular (IM) corticosteroid dose and/or hospitalization and/or emergency department (ED) visits. For participants on maintenance systemic corticosteroids, at least double the existing maintenance dose for at least 3 days is required. Percentage of participants with clinically significant exacerbation over time during the on-treatment period of Part C and 95% confidence interval were estimated using Kaplan-Meier estimates. Intent-to-Treat Population includes all randomized participants who received at least one dose of double-blind study medication within Part C.
Time Frame: Weeks 12, 24, 36 and 52
Population: Intent-to-Treat Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part C: Placebo | Part C: Mepolizumab 100mg SC
Number analyzed (Participants) | 151 | 144
Percentage of participants
  Week 12 | 31.8 [25.0 to 39.9] | 20.2 [14.5 to 27.7]
  Week 24 | 49.3 [41.5 to 57.6] | 32.3 [25.3 to 40.7]
  Week 36 | 56.0 [48.1 to 64.2] | 40.3 [32.8 to 48.9]
  Weeks 52 | 60.7 [52.7 to 68.8] | 47.1 [39.2 to 55.7]
Statistical Analysis 1: Comparison: Part C: Placebo vs Part C: Mepolizumab 100mg SC; Test type: Superiority; p = 0.004, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.45 to 0.86] — Treatment comparison between mepolizumab 100 mg SC and placebo using hazards ratio and 95% confidence interval has been presented

2. Secondary Outcome: Ratio to Baseline in Blood Eosinophil Count in Part C
Description: Blood samples were collected at specific time points to measure blood eosinophils level. Baseline was defined as the latest available assessment prior to first dose of double-blind treatment within Part C. Ratio to Baseline is defined as visit value divided by Baseline value and was analyzed using Mixed Model Repeated Measures with covariates of Baseline, region, exacerbations in the year prior to randomization (as an ordinal variable), Baseline maintenance oral corticosteroids (OCS) therapy (OCS versus no OCS), treatment and visit, plus interaction terms for visit by Baseline and visit by treatment group. The log transformation was applied to blood eosinophil counts prior to analysis. If a blood eosinophil count of zero was reported, a small value was added prior to log transforming the data. The dispersion measure used was log standard error.
Time Frame: Baseline and Weeks 12, 24, 36 and 52
Population: Intent-to-Treat Population. Only those participants available at the specified time points were analyzed for each treatment and represented as n=X in category titles
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Part C: Placebo | Part C: Mepolizumab 100mg SC
Number analyzed (Participants) | 121 | 120
Ratio
  Week 12, n=121, 120 | 6.03 (0.077) | 1.16 (0.078)
  Week 24, n= 79, 106: number analyzed (Participants) | 79 | 106
  Week 24, n= 79, 106 | 6.58 (0.095) | 1.03 (0.084)
  Week 36, n= 65, 99: number analyzed (Participants) | 65 | 99
  Week 36, n= 65, 99 | 6.48 (0.093) | 1.20 (0.079)
  Week 52, n=60, 92: number analyzed (Participants) | 60 | 92
  Week 52, n=60, 92 | 6.17 (0.091) | 1.00 (0.077)
Statistical Analysis 1: Comparison: Part C: Placebo vs Part C: Mepolizumab 100mg SC; Test type: Superiority; p < 0.001, Mixed model repeated measures; Ratio = 0.19, 95% CI 2-sided [0.15 to 0.24] — Treatment comparison between mepolizumab 100 mg SC and placebo using ratio of mepolizumab to placebo and its 95% confidence interval at Week 12 has been presented
Statistical Analysis 2: Comparison: Part C: Placebo vs Part C: Mepolizumab 100mg SC; Test type: Superiority; p < 0.001, Mixed model repeated measures; Ratio = 0.16, 95% CI 2-sided [0.12 to 0.20] — Treatment comparison between mepolizumab 100 mg SC and placebo using ratio of mepolizumab to placebo and its 95% confidence interval at Week 24 has been presented
Statistical Analysis 3: Comparison: Part C: Placebo vs Part C: Mepolizumab 100mg SC; Test type: Superiority; p < 0.001, Mixed model repeated measures; Ratio = 0.19, 95% CI 2-sided [0.15 to 0.24] — Treatment comparison between mepolizumab 100 mg SC and placebo using ratio of mepolizumab to placebo and its 95% confidence interval at Week 36 has been presented
Statistical Analysis 4: Comparison: Part C: Placebo vs Part C: Mepolizumab 100mg SC; Test type: Superiority; p < 0.001, Mixed model repeated measures; Ratio = 0.16, 95% CI 2-sided [0.13 to 0.20] — Treatment comparison between mepolizumab 100 mg SC and placebo using ratio of mepolizumab to placebo and its 95% confidence interval at Week 52 has been presented

3. Secondary Outcome: Percentage of Participants With 0.5 Point or More Increase in Asthma Control Questionnaire (ACQ)-5 Score From Baseline in Part C
Description: The ACQ-5 is a five-item, self-completed questionnaire. Five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response ranges from zero (no impairment/limitation) to six (total impairment/ limitation) scale. Increase in score of >= 0.5 units from Baseline indicates decrease in asthma control. Baseline is the latest available assessment prior to first dose of double-blind treatment within Part C. Percentage of participants with a 0.5 point or more increase in ACQ-5 score from Baseline over time during the on-treatment period of Part C and its 95% confidence interval were estimated using Kaplan-Meier estimates.
Time Frame: Baseline and Weeks 12, 24, 36 and 52
Population: Intent-to-Treat Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part C: Placebo | Part C: Mepolizumab 100mg SC
Number analyzed (Participants) | 151 | 144
Percentage of participants
  Week 12 | 44.5 [36.9 to 52.8] | 39.3 [31.8 to 47.8]
  Week 24 | 69.5 [61.6 to 77.1] | 49.3 [41.3 to 57.9]
  Week 36 | 74.9 [67.1 to 82.1] | 56.0 [47.8 to 64.6]
  Weeks 52 | 79.0 [71.3 to 85.7] | 63.1 [54.8 to 71.5]
Statistical Analysis 1: Comparison: Part C: Placebo vs Part C: Mepolizumab 100mg SC; Test type: Superiority; p = 0.005, Cox Proportional Hazards Model; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.49 to 0.88] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With Time to First Exacerbation Requiring Hospitalization or ED Visit in Part C
Description: Exacerbations of asthma requiring hospitalization or ED visit were assessed. The analysis was performed from Cox Proportional Hazards Model with covariates of treatment group, region, exacerbations in the year prior to randomization (as an ordinal variable) and Baseline maintenance OCS therapy (OCS versus no OCS). Percentage of participants with an exacerbation over time and its 95% confidence intervals were estimated using Kaplan-Meier estimates
Time Frame: Weeks 12, 24, 36 and 52
Population: Intent-to-Treat Population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part C: Placebo | Part C: Mepolizumab 100mg SC
Number analyzed (Participants) | 151 | 144
Percentage of participants
  Week 12 | 2.9 [1.1 to 7.5] | 2.8 [1.1 to 7.2]
  Week 24 | 5.7 [2.7 to 11.8] | 5.1 [2.4 to 10.3]
  Week 36 | 5.7 [2.7 to 11.8] | 5.9 [3.0 to 11.6]
  Weeks 52 | 5.7 [2.7 to 11.8] | 7.9 [4.3 to 14.3]
Statistical Analysis 1: Comparison: Part C: Placebo vs Part C: Mepolizumab 100mg SC; Test type: Superiority; p = 0.570, Cox Proportional Hazards Model; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.50 to 3.51] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) & Serious Adverse Events (SAEs) were collected for Part A/B: from first dose of OL mepolizumab in Parts A/B until the last dose of mepolizumab in Parts A/B (upto 132 weeks for Part A & upto 8 weeks for Part B); for Part C: from start of double blind treatment until the last dose of double-blind treatment (upto 52 weeks) & for Part D: from start of first dose of OL treatment in Part D until the last dose of OL treatment in Part D (upto 52 weeks post-randomization in Part C)
Description: AEs and SAEs were collected for As Treated Population which comprised of all participants who received at least one dose of open label mepolizumab for Parts A/B and Part D. Intent-to-Treat (ITT) Population was used for Part C which comprised of all randomized participants who received at least one dose of double-blind study medication. Combined data for parts A and B are presented since all par. received OL mepolizumab 100 mg SC.
Groups:
- Part C: Mepolizumab 100mg: Upon completion of the fixed run-in period, participants entered a double-blind study treatment and received continued mepolizumab 100 mg SC every 4 weeks up to 52 weeks. Participants who experienced a clinically significant asthma exacerbation were assessed by the investigator to determine if they could continue double-blind treatment or should instead enter OL mepolizumab 100 mg SC every 4 weeks for the remainder of the treatment period (up to 52 weeks post-randomization).
- Part D: Mepolizumab 100mg SC (Previous Mepolizumab): Participants who experienced a clinically significant asthma exacerbation were assessed by the investigator to determine if they could continue double-blind treatment or should instead enter OL mepolizumab 100 mg SC every 4 weeks for the remainder of the treatment period (up to 52 weeks post-randomization in Part C).
Arm/Group | Part A/B: Mepolizumab 100mg SC | Part C: Placebo | Part C: Mepolizumab 100mg | Part D: Mepolizumab 100mg SC (Previous Placebo) | Part D: Mepolizumab 100mg SC (Previous Mepolizumab)
All-Cause Mortality (participants affected / at risk) | 0/306 | 0/151 | 0/144 | 1/84 | 0/45
Serious Adverse Events (participants affected / at risk) | 7/306 | 10/151 | 9/144 | 10/84 | 4/45
Other Adverse Events (participants affected / at risk) | 14/306 | 69/151 | 82/144 | 44/84 | 32/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A/B: Mepolizumab 100mg SC (N=306) | Part C: Placebo (N=151) | Part C: Mepolizumab 100mg (N=144) | Part D: Mepolizumab 100mg SC (Previous Placebo) (N=84) | Part D: Mepolizumab 100mg SC (Previous Mepolizumab) (N=45)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (6) | 2 (2) | 4 (4) | 4 (6)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A/B: Mepolizumab 100mg SC (N=306) | Part C: Placebo (N=151) | Part C: Mepolizumab 100mg (N=144) | Part D: Mepolizumab 100mg SC (Previous Placebo) (N=84) | Part D: Mepolizumab 100mg SC (Previous Mepolizumab) (N=45)
Nasopharyngitis (Infections and infestations) | 14 (23) | 26 (44) | 27 (36) | 16 (22) | 9 (12)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 14 (18) | 12 (14) | 5 (5) | 3 (3)
Sinusitis (Infections and infestations) | 0 (0) | 9 (10) | 13 (14) | 7 (11) | 5 (8)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5) | 14 (14) | 7 (8) | 8 (13)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 2 (2) | 6 (11) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 5 (7) | 3 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 14 (16) | 10 (14) | 7 (7) | 4 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (12) | 6 (8) | 3 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 9 (11) | 9 (12) | 6 (7) | 4 (7)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/71/NCT02555371/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT02555371/SAP_001.pdf